CLINICAL TRIAL: NCT04039347
Title: A Phase III, Extension Clinical Trial to Demonstrate Efficacy and Safety of Liposomal Cyclosprine a Via the PARI Investigational EFlow® Device and SoC in Treating Bronchiolitis Obliterans in Patients Post Single or Double Lung Transplant
Brief Title: Extension Trial on Efficacy / Safety of L-CsA + SoC in Treating BOS in Post Single or Double Lung Transplant (BOSTON-3)
Acronym: BOSTON-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT - L-CsA - 303 - FU; 2019-002987-29 (EudraCT Number)
Record Dates: First submitted 2019-07-19; First posted 2019-07-31 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Bronchiolitis Obliterans; Obliterative Bronchiolitis; Bronchiolitis Obliterans Syndrome
Keywords: single and double transplant
MeSH Terms: conditions — Bronchiolitis Obliterans; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-CsA 5 mg plus Standard of Care (Experimental): L-CsA 5 mg twice daily plus Standard of Care for up to 144 weeks for patients post Single Lung Transplant
  Interventions: Drug: Liposomal Cyclosporine A 5 mg
- L-CsA 10 mg plus Standard of Care (Experimental): L-CsA 10 mg twice daily plus Standard of Care for up to 144 weeks for patients post Double Lung Transplant
  Interventions: Drug: Liposomal Cyclosporine A 10 mg

INTERVENTIONS:
Drug: Liposomal Cyclosporine A 5 mg — delivered via the PARI eFlow® device, which is a new technology of nebulizing liquid drugs with a perforated vibrating membrane resulting in an aerosol with a low ballistic momentum and a high percentage of droplets in a respirable size range of 3-5 μm
  Other Names: L-CsA
  Arms: L-CsA 5 mg plus Standard of Care
Drug: Liposomal Cyclosporine A 10 mg — delivered via the PARI eFlow® device, which is a new technology of nebulizing liquid drugs with a perforated vibrating membrane resulting in an aerosol with a low ballistic momentum and a high percentage of droplets in a respirable size range of 3-5 μm
  Other Names: L-CsA
  Arms: L-CsA 10 mg plus Standard of Care

SUMMARY:
The objective of the trial is to assess the long-term safety and efficacy of L-CsA plus Standard of Care (SoC) in the treatment of BOS in single (SLT) and double lung transplant (DLT) recipients.

DETAILED DESCRIPTION:
This is a Phase III, multicenter, open-label, extension clinical trial of L-CsA for the treatment of BOS.

Enrollment will be limited to patients who have completed 48 weeks participation in either the BT-L-CsA-301-SLT (BOSTON-1) or BT-L-CsA-302-DLT (BOSTON-2) trial. All patients in this clinical trial will receive L-CsA in addition to SoC, regardless of the randomization arm in prior trials.

IMP will be administered by BID inhalation (morning/evening) using the L-CsA eFlow. Patients who did not receive L-CsA in BOSTON-1 or BOSTON-2 must remain in the clinic for at least 4 hours for observation after the first inhalation. At all subsequent visits, one dose administered via inhalation will be monitored by the clinical trial center personnel. In case patients receiving L-CsA undergo the last visit for BOSTON-1 or BOSTON-2 (Visit 9) on the same day as for Visit 1 for BOSTON-3, they will take the first dose for Boston 3 in the evening of this day. This first dose will not be supervised by the site staff. Nebulization time per inhalation dose is approximately 6-10 minutes for the 5 mg dose and 9-13 minutes for the 10 mg dose. Inhalations will be performed BID approximately 12 hours apart through a mouthpiece by slow and deep respiration using the L-CsA eFlow. A high efficiency particulate air filter is used to prevent environmental contamination during exhalation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have completed all visits through the End of Treatment Visit in either BOSTON-1 or BOSTON-2, did not withdraw informed consent, and did not prematurely terminate study drug administration.
2. Patients should be on a three-drug maintenance regimen of immunosuppressive agents including tacrolimus or another CNI, a second agent such as but not limited to MMF or azathioprine, and a systemic corticosteroid such as prednisone.
3. Patients capable of understanding the purposes and risks of the clinical trial, who have given written informed consent and agree to comply with the clinical trial requirements/visit schedules, and who are capable of aerosol inhalation.
4. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to Visit 1 and must agree to use one of the methods of contraception listed in Appendix II through their End of Study Visit.

Exclusion Criteria:

1. Known hypersensitivity to L-CsA or to cyclosporine A.
2. Patients who experienced an AE related to study drug that led to permanent study drug discontinuation in BOSTON-1 or BOSTON-2.
3. Patients with new onset of malignancy while participating in BOSTON-1 or BOSTON-2, including post-transplant lymphoproliferative disorder, with the exception of treated, localized basal and squamous cell carcinomas.
4. Pregnant women or women who are unwilling to use appropriate birth control to avoid pregnancy through their End of Study Visit.
5. Women who are currently breastfeeding.
6. Receipt of an investigational drug, other than L-CsA, as part of a clinical trial within 4 weeks prior to Visit 1. This is defined as any treatment that is implemented under an Investigational New Drug (IND) or compassionate use.
7. Patients who are currently participating in an interventional clinical trial, other than BOSTON-1 or BOSTON-2.
8. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary procedures.
9. Any co-existing medical condition that in the Investigator's judgment will substantially increase the risk associated with the patient's participation in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean change in FEV1 from Baseline to Week 24 | Baseline to Week 24
  FEV1 is the Forced Expiratory Volume in One Second

SECONDARY OUTCOMES:
Mean change in FEV1 from Baseline to Week 48 | Baseline to Week 48
  FEV1 is the Forced Expiratory Volume in One Second
Mean change in FEV1 from Baseline to End of Study | Baseline to end of study, approximately 2 years
  FEV1 is the Forced Expiratory Volume in One Second
Mean change in FEV1/FVC from Baseline to Week 24 | Baseline to Week 24
  FEV1/FVC is the ratio between Forced Expiratory Volume in One Second and Forced Vital Capacity.
Mean change in FEV1/FVC from Baseline to Week 48 | Baseline to Week 48
  FEV1/FVC is the ratio between Forced Expiratory Volume in One Second and Forced Vital Capacity.
Time to Progression of BOS | Baseline to End of Study, approximately 2 years
  The Progression of BOS is defined as the earliest of:
  * Absolute decrease from baseline in FEV1 >/= 10% or >/= 200 mL and absolute decrease in FEV1/FVC of > 5%, OR
  * Change in BOS severity (according to criteria in Verleden 2019), OR
  * Re-transplantation, OR
  * Death from respiratory failure

OTHER OUTCOMES:
Adverse events | Baseline through end of study, approximately 2 years
  An untoward medical occurrence after exposure to a medicine, which is not necessarily caused by that medicine.
Acute tolerability of L-CsA as measured by change in FEV1 at 1 hour and 4 hours after first inhalation of L-CsA | First treatment with L-CsA
  Parameters reflecting acute tolerability of IMP are:
  * spirometry, before and 1 hour and 4 hours after inhalation of L-CsA at initial dosing.
  * cough, or
  * dyspnea.
Acute tolerability of L-CsA as measured by number of patients with treatment-related adverse events | Baseline through end of treatment, approximately 2 years
  Acute tolerability of L-CsA is measured by number of patients with treatment-related adverse events as assessed by CTCAE v5.0
Number of patients with treatment-related changes in hematology or serum chemistry parameters | Baseline through end of study participation, approximately 2 years
  Number of patients with treatment-related changes in hematology or serum chemistry parameters assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Paola R Castellani, MD, Study Director — Zambon SpA, Chief Medical Officer
Locations (37):
- United States (20):
  - Banner - University Medical Center, Phoenix, Arizona
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - UCSF, San Francisco, California
  - UCSF Center for Advanced Lung Disease, Stanford, California
  - University of Florida Dept of Pulmonary Medicine, Gainesville, Florida
  - Indiana University, Indianapolis, Indiana
  - UK Albert B. Chandler Hospital, Lexington, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
- Waehringer Guertel, Vienna, Austria
- Belgium (2):
  - Hôpital Erasme, Brussels
  - Universitair Ziekenhuis Leuven, Leuven
- Copenhagen University Hospital, Copenhagen, Denmark
- France (3):
  - Hopital Marie Lannelongue, Le Plessis-Robinson
  - CHU Hopital Nord, Marseille
  - Hopitaux Universitaires de Strasbourg, Strasbourg
- Germany (2):
  - Hannover Medical School, Hanover
  - LMU Klinikum Groshadern, Munich
- Rabin Medical Center, Petah Tikva, Israel
- Spain (5):
  - Complexo Hospitalario de A Coruna, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Puerta de Hierro - Unidad de Trasplante Pulmonar, Madrid
  - Hospital Marques de Valdecilla, Santander
  - Unidad de Trasplante Pulmonar del Hospital La Fe, Valencia
- United Kingdom (2):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - University of Manchester, Manchester

IPD SHARING:
Plan to Share IPD: No